CLINICAL TRIAL: NCT04350138
Title: A Phase II Randomized, Observer-Blind, Placebo-Controlled Study, to Assess the Efficacy of Meningococcal Group B Vaccine rMenB+OMV NZ (Bexsero) in Preventing Gonococcal Infection
Brief Title: Safety and Efficacy Study of Meningococcal Group B Vaccine rMenB+OMV NZ (Bexsero) to Prevent Gonococcal Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-0004; HHSN272201300012I
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-07-18

CONDITIONS: Gonococcal Infection
Keywords: Bexsero; Gonococcal infection; Meningococcal Group B Vaccine rMenB+OMV NZ; Observer-blind; Phase 2; Placebo-controlled study
MeSH Terms: conditions — Gonorrhea | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Bexsero vaccine will be administered as an intramuscular injection in 1 mL single-dose prefilled syringe in two doses with a two-month apart (at enrollment/Visit 1 and Visit 3). N=1100.
  Interventions: Biological: Meningococcal Group B Vaccine
- Group 2 (Placebo Comparator): Placebo will be administered as an intramuscular injection in single-dose prefilled syringe in two doses with a two-month apart (at enrollment/Visit 1 and Visit 3). N=1100.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Meningococcal Group B Vaccine — A combination vaccine consisting of rMenB and OMV NZ.
  Arms: Group 1
Other: Placebo — 150mM sodium chloride (0.9% saline solution).
  Arms: Group 2

SUMMARY:
This is a Phase II, randomized, observer-blind, placebo-controlled, multi-site trial of the FDA licensed rMenB+OMV NZ vaccine, Bexsero. The targeted study population is men and women 18-50 years of age who are disproportionately vulnerable to N. gonorrhoeae infection. Approximately 2,200 participants are expected to be enrolled to achieve at least 202 primary endpoints in the Per Protocol Population. Data will be collected in an observer-blind manner. Study product recipients and study staff responsible for the evaluation of any study endpoint will be unaware of whether Bexsero or placebo were administered. The duration of the study for participants who are enrolled and randomized will be approximately 16 months. Study participation is expected to be completed in approximately 36 months. The primary objective of the study is to demonstrate efficacy of Bexsero in prevention of urogenital and/or anorectal gonococcal infection.

DETAILED DESCRIPTION:
This is a Phase II, randomized, observer-blind, placebo-controlled, multi-site trial of the FDA licensed rMenB+OMV NZ vaccine, Bexsero. The targeted study population is men and women 18-50 years of age who are disproportionately vulnerable to N. gonorrhoeae infection. Approximately 2,200 participants are expected to be enrolled to achieve at least 202 primary endpoints in the Per Protocol Population. Data will be collected in an observer-blind manner. Study product recipients and study staff responsible for the evaluation of any study endpoint will be unaware of whether Bexsero or placebo were administered. Participants who consent to screening will have baseline clinical information collected at Visit 0, Screening (Day -14 [Window -45 to -7]). This information will consist of medical history, concomitant medications, physical exam, sexual history, and clinical and laboratory findings. Participants will undergo a physical exam and have blood drawn to establish baseline laboratory values for safety assessment. Urine or a vaginal swab, and a rectal swab will be collected for Nucleic Acid Amplification Test (NAAT) for gonorrhea and chlamydia. A pharyngeal swab will be collected for NAAT testing of gonorrhea. At the enrollment visit, Visit 1, participants who test negative for gonorrhea and who otherwise qualify will be enrolled and randomized in a 1:1 ratio to receive the initial intramuscular (IM) dose of study product. A phone call, Visit 2, will be held approximately 30 days after the initial study product dose was received and will be conducted with all participants to assess for safety events in the interim. At Visit 3, the participant will receive the second dose of study product. Visit 4 will be held 1 month after second dose. At 3-month intervals, through the final study follow-up visit, participants will have clinic study visits, Visit 5 thru Visit 8. The duration of the study for participants who are enrolled and randomized will be approximately 16 months. For those not enrolled, participation could end at their Visit 0, Screening; post Visit 0, Screening based on NAAT test results; or Visit 1, Enrollment. Study participation is expected to be completed in approximately 36 months. The primary objective of the study is to demonstrate efficacy of Bexsero in prevention of urogenital and/or anorectal gonococcal infection. The secondary objectives are to estimate efficacy of Bexsero in prevention of overall gonococcal infection and by anatomical site (urogenital, anorectal or pharyngeal) and to assess safety of Bexsero.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 50 years of age inclusive on the day of enrollment;
2. If female, participant must be of non-childbearing potential* or has a negative pregnancy test prior to each vaccination**.

   *Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopausal (no menses for at least 12 months);

   **Note: Although contraceptive methods are not mandated since Bexsero is a marketed product and will be used according to the label, it is anticipated that contraceptive counselling will be provided according to local standard of care.
3. Participant is in good health as determined by past medical history, medication use, and targeted physical examination (including vital signs), in opinion of investigator or their delegate;
4. Has provided signed informed consent;
5. Willing and likely to comply with the trial procedures;
6. Is prepared to grant authorized persons access to the study's medical records.

Exclusion Criteria:

1. Previous receipt of a Meningococcal Group B vaccine;
2. Gonorrhea or chlamydia infection identified by a positive nucleic acid amplification test (NAAT) within 14 days prior to randomization;
3. Receipt of antibiotics active against N. gonorrhoeae in the prior 14 days, including oral or parenteral antibiotics;
4. Progressive, unstable, or uncontrolled disease including but not limited to cardiac, hepatic, renal, immunological, neurological or psychiatric conditions;
5. Use of any investigational drug (with the exception of an authorized or approved COVID-19 vaccine) within 30 days prior to enrollment, or planned/anticipated use during study participation;
6. Has received or plans to receive a live vaccine within +/- 30 days, an inactive vaccine within +/- 14 days, or an influenza vaccine within +/- 7 days from receipt of study product;*

   *Authorized or approved, inactivated COVID-19 vaccines may be given more than 7 days +/- receipt of study product for all study participants.
7. Currently receiving immunosuppressive agent or systemic corticosteroid (dose >/=5 mg/day of prednisone) for > 14 consecutive days within 90 days prior to enrollment*;

   *Topical or inhaled steroids allowed, unless applied to study project injection site.
8. Has received antineoplastic, or radiotherapy within 90 days prior to enrollment;
9. Has received immunoglobulins and/or any blood products within 180 days prior to enrollment;
10. Known or confirmed hypersensitivity to any of the vaccine constituents, medical products, or medical equipment whose use is foreseen in this study;
11. HIV-infected participants with CD4 cell count < 300 cells/mm3 in the last year;
12. Has a condition which in the opinion of the investigator is not suitable for intramuscular vaccination, blood draws, or participation in the trial;
13. Participant is breastfeeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2606 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants diagnosed with urogenital or anorectal gonococcal infection post second vaccination | Day 91 to Day 451
  Confirmed by Nucleic Acid Amplification Test (NAAT).

SECONDARY OUTCOMES:
Number of participants diagnosed with urogenital, anorectal, or pharyngeal gonococcal infection post second vaccination | Day 91 to Day 451
  Confirmed by Nucleic Acid Amplification Test (NAAT).
Proportion of participants that experience at least one adverse event (AE) that results in withdrawal from study | Day 1 to Day 451
  Disease or medical condition, or new clinical finding(s) for which continued participation, in the opinion of the investigator might compromise the safety of the participant, interfere with the participant's successful completion of this study, or interfere with the evaluation of study endpoints.
Proportion of participants that experience at least one adverse event of special interest (AESI) | Day 1 to Day 451
  Adverse Event of Special Interest (AESI) are specific to the protocol: Arthritis, Potential immune-mediated diseases (pIMD).
Proportion of participants that experience at least one serious adverse event (SAE) | Day 1 to Day 451
Proportion of participants with at least one medically attended adverse event (MAAE) | Day 1 to Day 451

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - SFDPH Bridge HIV Center, San Francisco, California
  - Emory University School of Medicine - The Ponce de Leon Center, Atlanta, Georgia
  - Emory University Hospital Midtown - Emory Clinic Infectious Diseases, Atlanta, Georgia
  - University of Illinois at Chicago College of Medicine - Division of Infectious Diseases, Chicago, Illinois
  - LSU - CrescentCare Sexual Health Center, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Harlem Prevention Center, Columbia University, Mailman School of Public Health, New York, New York
  - University of Pennsylvania HIV/AIDS Prevention Research Division, Philadelphia, Pennsylvania
- Malawi Clinical Research Site, Lilongwe, Lilongwe, Central Region, Malawi
- Thailand (2):
  - The Thai Red Cross AIDS Research Centre, Bangkok
  - Armed Forces Research Institute of Medical Sciences - Royal Thai Army Clinical Research Center, Bangkok